CLINICAL TRIAL: NCT04822480
Title: A Telehealth Diabetes Prevention Program in an Academic Medical Center Setting: Hybrid Type III Trial
Brief Title: Evaluation of a Telehealth DPP With Medicare Patients at the University of Mississippi Medical Center
Status: Active, not recruiting | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: American Medical Association (Other); Mississippi State Department of Health (Other Government)
Responsible Party: Principal Investigator, Abigail Gamble, Assistant Professor of Preventive Medicine and Population Health Science, University of Mississippi Medical Center
Other Study IDs: 2020V0327
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: PreDiabetes; Prediabetic State
Keywords: diabetes prevention
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DPP Patients: UMMC Patients with prediabetes or risk for diabetes based on risk parameters referred to and enrolled in the DPP.
  Interventions: Behavioral: Diabetes Prevention Program (DPP)
- Non-DPP Patients: Control matched UMMC patients with prediabetes or risk for diabetes based on risk parameters not enrolled in the DPP.

INTERVENTIONS:
Behavioral: Diabetes Prevention Program (DPP) — Individuals with prediabetes can mitigate the risks and costs of diabetes by taking preventative action, such as participation in a National Diabetes Prevention Program (DPP). The DPP began as a multisite randomized controlled trial demonstrating the effectiveness and cost-benefit of a 12-month intensive lifestyle intervention over pharmaceutical treatment for preventing or delaying diabetes among prediabetic participants. In 2010, Congress authorized the Centers for Disease Control and Prevention to lead the dissemination of the DPP as a targeted approach (high risk populations) and population-based strategy to reduce the incidence of diabetes and diabetes-related healthcare costs. The goal is to achieve modest weight loss (7%) by developing and implementing behavior change skills resulting in lifestyle modifications such as physical activity (150 minutes per week) and dietary and nutritional practices.
  Groups: DPP Patients

SUMMARY:
The National Diabetes Prevention Program (DPP) is an evidence-based, 12-month lifestyle change program to prevent or delay the onset of type 2 diabetes mellitus (herein referred to as 'diabetes') among adults with prediabetes. The Department of Preventive Medicine, University of Mississippi Medical Center (UMMC), in partnership with the American Medical Association, is collaborating to develop and implement the DPP as a clinical service for UMMC patients beginning in September 2020. We aim to recruit 245 patients per year over 3 years. Because this is the first attempt to develop and implement the DPP as a clinical service at the UMMC, we are proposing to conduct a comprehensive process, outcome, impact and return on investment evaluation. An effectiveness-implementation hybrid research design will be used to (1) evaluate a multifaceted implementation strategy and the effectiveness and impact of the DPP delivered using telehealth by UMMC's Department of Preventive Medicine; (2) conduct an analysis on medical expenditures among those who participate in a DPP to measure net savings and return on investment (ROI) relative to non-participants; (3) conduct a longitudinal cohort analysis to assess incidence of diabetes and changes in body composition, biomarkers, and psycho-social behavioral constructs among those who participate in a DPP relative to those who do not.

The findings from this comprehensive research evaluation will be used to (1) improve clinical operations and implementation; (2) demonstrate the cost benefit of the DPP as a clinical service for patients with diabetes risk; and (3) provide empirical support for delivering the DPP via different modalities including telehealth to reduce risk and improve health outcomes among patients.

DETAILED DESCRIPTION:
The purpose of this research is to: (1) Evaluate a multifaceted implementation strategy for the uptake of a remote DPP by UMMC's Department of Preventive Medicine. (2) Conduct an analysis on medical expenditures among those who participate in a DPP to measure net savings and ROI relative to non-participants. (3) Conduct a longitudinal cohort analysis to assess incidence of diabetes, body composition, biomarkers, and psycho-social behavioral constructs among those who participate in a DPP relative to those who do not. Study methods are described below according to each of three specific aims.

Aim 1: Conduct a concurrent implementation and effectiveness evaluation of the DPP in a clinical care setting for patients with prediabetes (n=245). An effectiveness-implementation hybrid type III research design will be used to conduct a non-randomized trial with 245 of patients with prediabetes over a three year recruitment period, while employing an iterative process evaluation to explore the complex processes, dynamic context and organizational influences on implementation. The RE-AIM framework will guide the implementation and effectiveness evaluation including measures of Reach, Effectiveness, Adoption, Implementation and Maintenance. Multiple data sources and data types will be used to assess barriers and facilitators that affect the RE-AIM domains, as well as fidelity, costs, patient satisfaction and physician burnout.

Aim 2: Utilize claims and encounters data to measure medical expenditures for patients with prediabetes, and determine spending differentials among DPP participants compared with non-DPP participants. Track trends in per capita medical expenditures for among a panel of case (DPP participant) and control (Non-DPP participant) subjects. To compare variations in spending, the differences in the arithmetic means, compound annual growth rates, and propensity score matching models will be implemented to compare case and control subjects. The study may also look at those with prediabetes that are later diagnosed with diabetes and individuals with prediabetes who are not later diagnosed with the condition. These estimates of spending differentials and evidence of DPP participation and engagement rates will help to further enhance the algorithm to estimate the potential cost savings and ROI if diabetes is prevented or delayed in the at-risk population who participate in the DPP.

Aim 3: Assess the longitudinal effect of the DPP on participant changes in cardiovascular disease risk including anthropometric and clinical biomarker and psychosocial health outcomes (N=245). A prospective, repeated measures, experimental cohort design will be used to determine the long-term impact of the DPP on diabetes incidence and cardiovascular disease risk among DPP patient participants.

ELIGIBILITY:
Inclusion Criteria:

* UMMC patient within the previous 3-years (at least one UMMC clinical visit within the previous 3-years)
* ≥ 18 years AND
* Clinical diagnosis for prediabetes (R73.03)

OR any of the following combinations:

* BMI ≥25 (non-Asian) OR
* BMI ≥23 (Asian) AND
* HbA1c 5.7 - 6.4 percent within the past 12-months OR
* Fasting plasma glucose 110 - 125 mg/dL within the past 12-months OR
* 2-hour plasma glucose 140 - 199 mg/dL within the past 12-months

Exclusion Criteria:

* Pregnant or planning to become pregnant within the next 12 months
* <18 years
* Primary or secondary diagnosis of diabetes mellitus (all codes with prefix of 250 and 249) and other conditions associated with diabetes (357.2, all codes with prefix 362, 366.41, and all codes with prefix 648).
* End stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mississippi consistently has among the highest rates of diabetes (14.3%) and prediabetes (36.5%) nationally and is the only state where every county (82 counties) are represented in the Diabetes Belt, a geographic region of the U.S. where the prevalence of diagnosed diabetes is highest. Mississippi has the fourth largest rural population (51.2%) and the highest state percent Black (37.8%) population in the U.S., and has persistently high rates of poverty (20.8%).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Type 2 diabetes mellitus diagnosis | Change diabetes diagnosis from baseline to 6-months in DPP compared with non-DPP patients
  Diabetes diagnosis extracted via electronic health record; all codes with prefix of 250 and 249
Type 2 diabetes mellitus diagnosis | Change diabetes diagnosis from baseline to 12-months in DPP compared with non-DPP patients
  Diabetes diagnosis extracted via electronic health record; all codes with prefix of 250 and 249
Type 2 diabetes mellitus diagnosis | Change diabetes diagnosis from baseline to 18-months in DPP compared with non-DPP patients
  Diabetes diagnosis extracted via electronic health record; all codes with prefix of 250 and 249
Type 2 diabetes mellitus diagnosis | Change diabetes diagnosis from baseline to 24-months in DPP compared with non-DPP patients
  Diabetes diagnosis extracted via electronic health record; all codes with prefix of 250 and 249
Type 2 diabetes mellitus diagnosis | Change diabetes diagnosis from baseline to 30-months in DPP compared with non-DPP patients
  Diabetes diagnosis extracted via electronic health record; all codes with prefix of 250 and 249
Type 2 diabetes mellitus diagnosis | Change diabetes diagnosis from baseline to 36-months in DPP compared with non-DPP patients
  Diabetes diagnosis extracted via electronic health record; all codes with prefix of 250 and 249
Hemoglobin A1c | Change in HbA1c from baseline to 6-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Hemoglobin A1c | Change in HbA1c from baseline to 12-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Hemoglobin A1c | Change in HbA1c from baseline to 18-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Hemoglobin A1c | Change in HbA1c from baseline to 24-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Hemoglobin A1c | Change in HbA1c from baseline to 30-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Hemoglobin A1c | Change in HbA1c from baseline to 36-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Fasting plasma glucose | Change in fasting plasma glucose from baseline to 6-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Fasting plasma glucose | Change in fasting plasma glucose from baseline to 12-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Fasting plasma glucose | Change in fasting plasma glucose from baseline to 18-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Fasting plasma glucose | Change in fasting plasma glucose from baseline to 24-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Fasting plasma glucose | Change in fasting plasma glucose from baseline to 30-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Fasting plasma glucose | Change in fasting plasma glucose from baseline to 36-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
2-hour plasma glucose | Change in 2-hour plasma glucose from baseline to 6-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
2-hour plasma glucose | Change in 2-hour plasma glucose from baseline to 12-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
2-hour plasma glucose | Change in 2-hour plasma glucose from baseline to 18-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
2-hour plasma glucose | Change in 2-hour plasma glucose from baseline to 24-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
2-hour plasma glucose | Change in 2-hour plasma glucose from baseline to 30-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
2-hour plasma glucose | Change in 2-hour plasma glucose from baseline to 36-months in DPP compared with non-DPP patients
  Lab values extracted from electronic health record
Medical encounters | Number of medical encounters between baseline and 6-months in DPP compared with non-DPP patients
  Extracted from electronic health record
Medical encounters | Number of medical encounters between baseline and 12-months in DPP compared with non-DPP patients
  Extracted from electronic health record
Medical encounters | Number of medical encounters between baseline and 18-months in DPP compared with non-DPP patients
  Extracted from electronic health record
Medical encounters | Number of medical encounters between baseline and 24-months in DPP compared with non-DPP patients
  Extracted from electronic health record
Medical encounters | Number of medical encounters between baseline and 30-months in DPP compared with non-DPP patients
  Extracted from electronic health record
Medical encounters | Number of medical encounters between baseline and 36-months in DPP compared with non-DPP patients
  Extracted from electronic health record
Medical expenditures | Medical expenditures from baseline to 6-months in DPP compared with non-DPP patients
  Total dollar amount billed per encounter extracted from electronic health record
Medical expenditures | Medical expenditures from baseline to 12-months in DPP compared with non-DPP patients
  Total dollar amount billed per encounter extracted from electronic health record
Medical expenditures | Medical expenditures from baseline to 18-months in DPP compared with non-DPP patients
  Total dollar amount billed per encounter extracted from electronic health record
Medical expenditures | Medical expenditures from baseline to 24-months in DPP compared with non-DPP patients
  Total dollar amount billed per encounter extracted from electronic health record
Medical expenditures | Medical expenditures from baseline to 30-months in DPP compared with non-DPP patients
  Total dollar amount billed per encounter extracted from electronic health record
Medical expenditures | Medical expenditures from baseline to 36-months in DPP compared with non-DPP patients
  Total dollar amount billed per encounter extracted from electronic health record

SECONDARY OUTCOMES:
Body weight | Change in body weight from baseline to 6-months
  Total body weight measured using Seca mBCA 554
Body weight | Change in body weight from baseline to 12-months
  Total body weight measured using Seca mBCA 554
Body weight | Change in body weight from baseline to 24-months
  Total body weight measured using Seca mBCA 554
Body weight | Change in body weight from baseline to 36-months
  Total body weight measured using Seca mBCA 554
Fat mass | Change in fat mass from baseline to 6-months
  Total body fat mass measured using Seca mBCA 554; bioimpedance analysis
Fat mass | Change in fat mass from baseline to 12-months
  Total body fat mass measured using Seca mBCA 554; bioimpedance analysis
Fat mass | Change in fat mass from baseline to 24-months
  Total body fat mass measured using Seca mBCA 554; bioimpedance analysis
Fat mass | Change in fat mass from baseline to 36-months
  Total body fat mass measured using Seca mBCA 554; bioimpedance analysis
Visceral fat | Change in visceral fat from baseline to 6-months
  Visceral fat measured using Seca mBCA 554; bioimpedance analysis
Visceral fat | Change in visceral fat from baseline to 12-months
  Visceral fat measured using Seca mBCA 554; bioimpedance analysis
Visceral fat | Change in visceral fat from baseline to 24-months
  Visceral fat measured using Seca mBCA 554; bioimpedance analysis
Visceral fat | Change in visceral fat from baseline to 36-months
  Visceral fat measured using Seca mBCA 554; bioimpedance analysis
Skeletal muscle mass | Change in skeletal muscle mass from baseline to 6-months
  Total body skeletal muscle mass measured using Seca mBCA 554; bioimpedance analysis
Skeletal muscle mass | Change in skeletal muscle mass from baseline to 12-months
  Total body skeletal muscle mass measured using Seca mBCA 554; bioimpedance analysis
Skeletal muscle mass | Change in skeletal muscle mass from baseline to 24-months
  Total body skeletal muscle mass measured using Seca mBCA 554; bioimpedance analysis
Skeletal muscle mass | Change in skeletal muscle mass from baseline to 36-months
  Total body skeletal muscle mass measured using Seca mBCA 554; bioimpedance analysis
Waist circumference | Change in waist circumference from baseline to 6-months
  Measures using Seca 203 circumference measuring tape
Waist circumference | Change in waist circumference from baseline to 12-months
  Measures using Seca 203 circumference measuring tape
Waist circumference | Change in waist circumference from baseline to 24-months
  Measures using Seca 203 circumference measuring tape
Waist circumference | Change in waist circumference from baseline to 36-months
  Measures using Seca 203 circumference measuring tape
Systolic blood pressure | Change in systolic blood pressure from baseline to 6-months
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Systolic blood pressure | Change in systolic blood pressure from baseline to 12-months
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Systolic blood pressure | Change in systolic blood pressure from baseline to 24-months
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Systolic blood pressure | Change in systolic blood pressure from baseline to 36-months
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Diastolic blood pressure | Change in diastolic blood pressure from baseline to 6-months
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Diastolic blood pressure | Change in diastolic blood pressure from baseline to 12-months
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Diastolic blood pressure | Change in diastolic blood pressure from baseline to 24-months
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Diastolic blood pressure | Change in diastolic blood pressure from baseline to 36-months
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Resting heart rate | Change in resting heart rate from baseline to 6-months
  Welch Allyn blood pressure unit.
Resting heart rate | Change in resting heart rate from baseline to 12-months
  Welch Allyn blood pressure unit.
Resting heart rate | Change in resting heart rate from baseline to 24-months
  Welch Allyn blood pressure unit.
Resting heart rate | Change in resting heart rate from baseline to 36-months
  Welch Allyn blood pressure unit.
Total cholesterol | Change in total cholesterol from baseline to 6-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
Total cholesterol | Change in total cholesterol from baseline to 12-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
Total cholesterol | Change in total cholesterol from baseline to 24-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
Total cholesterol | Change in total cholesterol from baseline to 36-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
HDL cholesterol | Change in HDL cholesterol from baseline to 6-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
HDL cholesterol | Change in HDL cholesterol from baseline to 12-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
HDL cholesterol | Change in HDL cholesterol from baseline to 24-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
HDL cholesterol | Change in HDL cholesterol from baseline to 36-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
Triglycerides | Change in triglycerides from baseline to 6-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
Triglycerides | Change in triglycerides from baseline to 12-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
Triglycerides | Change in triglycerides from baseline to 24-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
Triglycerides | Change in triglycerides from baseline to 36-months
  PTS Diagnostics CardioChek Plus analyzer; point of care finger stick to obtain 40 μL blood
Hemoglobin A1c (point of care) | Change in HbA1c from baseline to 6-months
  A1CNOW+ System for reliable point-of-care HbA1c measurement; non-fasting 5 μL blood
Hemoglobin A1c (point of care) | Change in HbA1c from baseline to 12-months
  A1CNOW+ System for reliable point-of-care HbA1c measurement; non-fasting 5 μL blood
Hemoglobin A1c (point of care) | Change in HbA1c from baseline to 24-months
  A1CNOW+ System for reliable point-of-care HbA1c measurement; non-fasting 5 μL blood
Hemoglobin A1c (point of care) | Change in HbA1c from baseline to 36-months
  A1CNOW+ System for reliable point-of-care HbA1c measurement; non-fasting 5 μL blood
Self-efficacy for weight loss and maintenance | Change in self-efficacy from baseline to 6-months
  Weight self-efficacy lifestyle questionnaire; 20 items using a 10-point Likert scale; higher mean score indicates higher self-efficacy; Clark et al., 1991
Self-efficacy for weight loss and maintenance | Change in self-efficacy from baseline to 12-months
  Weight self-efficacy lifestyle questionnaire; 20 items using a 10-point Likert scale; higher mean score indicates higher self-efficacy; Clark et al., 1991
Self-efficacy for weight loss and maintenance | Change in self-efficacy from baseline to 24-months
  Weight self-efficacy lifestyle questionnaire; 20 items using a 10-point Likert scale; higher mean score indicates higher self-efficacy; Clark et al., 1991
Self-efficacy for weight loss and maintenance | Change in self-efficacy from baseline to 36-months
  Weight self-efficacy lifestyle questionnaire; 20 items using a 10-point Likert scale; higher mean score indicates higher self-efficacy; Clark et al., 1991
Readiness to change, stage of change | Change in stage of change from baseline to 6-months
  Stages of Change in Overweight and Obese People questionnaire (S-weight); 1-item with 5 distinct and mutually exclusive responses to measure stage of change; Andres et al., 2009
Readiness to change, stage of change | Change in stage of change from baseline to 12-months
  Stages of Change in Overweight and Obese People questionnaire (S-weight); 1-item with 5 distinct and mutually exclusive responses to measure stage of change; Andres et al., 2009
Readiness to change, stage of change | Change in stage of change from baseline to 24-months
  Stages of Change in Overweight and Obese People questionnaire (S-weight); 1-item with 5 distinct and mutually exclusive responses to measure stage of change; Andres et al., 2009
Readiness to change, stage of change | Change in stage of change from baseline to 36-months
  Stages of Change in Overweight and Obese People questionnaire (S-weight); 1-item with 5 distinct and mutually exclusive responses to measure stage of change; Andres et al., 2009
Readiness to change, processes of change | Change in processes of change from baseline to 6-months
  Processes of Change in Overweight and Obese People questionnaire (P-weight); 34 items; 5-point Likert scale from Strongly Disagree to Strongly Agree where higher mean score indicates higher use of respective process; four processes include emotional re-evaluation, weight consequences evaluation, supporting relationships, and weight management actions across 4 processes of change; Andres et al., 2011
Readiness to change, processes of change | Change in processes of change from baseline to 12-months
  Processes of Change in Overweight and Obese People questionnaire (P-weight); 34 items; 5-point Likert scale from Strongly Disagree to Strongly Agree where higher mean score indicates higher use of respective process; four processes include emotional re-evaluation, weight consequences evaluation, supporting relationships, and weight management actions across 4 processes of change; Andres et al., 2011
Readiness to change, processes of change | Change in processes of change from baseline to 24-months
  Processes of Change in Overweight and Obese People questionnaire (P-weight); 34 items; 5-point Likert scale from Strongly Disagree to Strongly Agree where higher mean score indicates higher use of respective process; four processes include emotional re-evaluation, weight consequences evaluation, supporting relationships, and weight management actions across 4 processes of change; Andres et al., 2011
Readiness to change, processes of change | Change in processes of change from baseline to 36-months
  Processes of Change in Overweight and Obese People questionnaire (P-weight); 34 items; 5-point Likert scale from Strongly Disagree to Strongly Agree where higher mean score indicates higher use of respective process; four processes include emotional re-evaluation, weight consequences evaluation, supporting relationships, and weight management actions across 4 processes of change; Andres et al., 2011
Decisional balance | Change in decisional balance from baseline to 6-months
  Decisional balance inventory; 20 items using 5-point Likert scale to identify cognitive and emotional pros and cons to making intentional changes for weight loss and maintenance (Not Important At All to Extremely Important); higher mean scores for subscales (Pros; Pro-Con) would indicate higher intention; O'Connell and Velicer, 1988
Decisional balance | Change in decisional balance from baseline to 12-months
  Decisional balance inventory; 20 items using 5-point Likert scale to identify cognitive and emotional pros and cons to making intentional changes for weight loss and maintenance (Not Important At All to Extremely Important); higher mean scores for subscales (Pros; Pro-Con) would indicate higher intention; O'Connell and Velicer, 1988
Decisional balance | Change in decisional balance from baseline to 24-months
  Decisional balance inventory; 20 items using 5-point Likert scale to identify cognitive and emotional pros and cons to making intentional changes for weight loss and maintenance (Not Important At All to Extremely Important); higher mean scores for subscales (Pros; Pro-Con) would indicate higher intention; O'Connell and Velicer, 1988
Decisional balance | Change in decisional balance from baseline to 36-months
  Decisional balance inventory; 20 items using 5-point Likert scale to identify cognitive and emotional pros and cons to making intentional changes for weight loss and maintenance (Not Important At All to Extremely Important); higher mean scores for subscales (Pros; Pro-Con) would indicate higher intention; O'Connell and Velicer, 1988
Self-efficacy for overcoming barriers to physical activity and healthy eating | Change in barrier self-efficacy from baseline to 6-months
  Self-efficacy for overcoming barriers to physical activity and diet; 10 items using a 4-point Likert scale from Very Uncertain to Very Certain or Not True At All to Exactly True; higher mean score (20 to 80) indicated greater self-efficacy; Huttunen-Lenz et al., 2018
Self-efficacy for overcoming barriers to physical activity and healthy eating | Change in barrier self-efficacy from baseline to 12-months
  Self-efficacy for overcoming barriers to physical activity and diet; 10 items using a 4-point Likert scale from Very Uncertain to Very Certain or Not True At All to Exactly True; higher mean score (20 to 80) indicated greater self-efficacy; Huttunen-Lenz et al., 2018
Self-efficacy for overcoming barriers to physical activity and healthy eating | Change in barrier self-efficacy from baseline to 24-months
  Self-efficacy for overcoming barriers to physical activity and diet; 10 items using a 4-point Likert scale from Very Uncertain to Very Certain or Not True At All to Exactly True; higher mean score (20 to 80) indicated greater self-efficacy; Huttunen-Lenz et al., 2018
Self-efficacy for overcoming barriers to physical activity and healthy eating | Change in barrier self-efficacy from baseline to 36-months
  Self-efficacy for overcoming barriers to physical activity and diet; 10 items using a 4-point Likert scale from Very Uncertain to Very Certain or Not True At All to Exactly True; higher mean score (20 to 80) indicated greater self-efficacy; Huttunen-Lenz et al., 2018
Self-regulation of eating behaviors | Change in self-regulation of eating behaviors from baseline to 6-months
  Self-regulation of Eating Behavior Questionnaire; 5 items using a 5-point Likert scale; mean score <2.8, 2.8 - 3.6, >3.6 correspond to low, medium and high self-regulation, respectively; Kliemann et al., 2016
Self-regulation of eating behaviors | Change in self-regulation of eating behaviors from baseline to 12-months
  Self-regulation of Eating Behavior Questionnaire; 5 items using a 5-point Likert scale; mean score <2.8, 2.8 - 3.6, >3.6 correspond to low, medium and high self-regulation, respectively; Kliemann et al., 2016
Self-regulation of eating behaviors | Change in self-regulation of eating behaviors from baseline to 24-months
  Self-regulation of Eating Behavior Questionnaire; 5 items using a 5-point Likert scale; mean score <2.8, 2.8 - 3.6, >3.6 correspond to low, medium and high self-regulation, respectively; Kliemann et al., 2016
Self-regulation of eating behaviors | Change in self-regulation of eating behaviors from baseline to 36-months
  Self-regulation of Eating Behavior Questionnaire; 5 items using a 5-point Likert scale; mean score <2.8, 2.8 - 3.6, >3.6 correspond to low, medium and high self-regulation, respectively; Kliemann et al., 2016
Self-regulation of physical activity - goals | Change in self-regulation of physical activity goals from baseline to 6-months
  Exercise goal-setting scale; 10 items using 5-point Likert scale from Does Not Describe Me (0) to Describes Me Completely (4); higher mean score reflects greater self-regulation Rovniak et al., 2002
Self-regulation of physical activity - goals | Change in self-regulation of physical activity goals from baseline to 12-months
  Exercise goal-setting scale; 10 items using 5-point Likert scale from Does Not Describe Me (0) to Describes Me Completely (4); higher mean score reflects greater self-regulation Rovniak et al., 2002
Self-regulation of physical activity - goals | Change in self-regulation of physical activity goals from baseline to 24-months
  Exercise goal-setting scale; 10 items using 5-point Likert scale from Does Not Describe Me (0) to Describes Me Completely (4); higher mean score reflects greater self-regulation Rovniak et al., 2002
Self-regulation of physical activity - goals | Change in self-regulation of physical activity goals from baseline to 36-months
  Exercise goal-setting scale; 10 items using 5-point Likert scale from Does Not Exercise goal-setting scale; 10 items using 5-point Likert scale from Does Not Describe Me (0) to Describes Me Completely (4); higher mean score reflects greater self-regulation Rovniak et al., 2002
Self-regulation of physical activity - planning | Change in self-regulation of physical activity planning from baseline to 6-months
  Exercise planning and scheduling scale; 10 items using 5-point Likert scale from Does Not Describe Me (0) to Describes Me Completely (4); higher mean score reflects greater self-regulation Rovniak et al., 2002
Self-regulation of physical activity - planning | Change in self-regulation of physical activity planning from baseline to 12-months
  Exercise planning and scheduling scale; 10 items using 5-point Likert scale from Does Not Describe Me (0) to Describes Me Completely (4); higher mean score reflects greater self-regulation Rovniak et al., 2002
Self-regulation of physical activity - planning | Change in self-regulation of physical activity planning from baseline to 24-months
  Exercise planning and scheduling scale; 10 items using 5-point Likert scale from Does Not Describe Me (0) to Describes Me Completely (4); higher mean score reflects greater self-regulation Rovniak et al., 2002
Self-regulation of physical activity - planning | Change in self-regulation of physical activity planning from baseline to 36-months
  Exercise planning and scheduling scale; 10 items using 5-point Likert scale from Does Not Describe Me (0) to Describes Me Completely (4); higher mean score reflects greater self-regulation Rovniak et al., 2002
Social support from friends - eating | Change in social support from baseline to 6-months
  Friend social support for healthy eating scale; 10 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from friends - eating | Change in social support from baseline to 12-months
  Friend social support for healthy eating scale; 10 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from friends - eating | Change in social support from baseline to 24-months
  Friend social support for healthy eating scale; 10 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from friends - eating | Change in social support from baseline to 36-months
  Friend social support for healthy eating scale; 10 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from family - eating | Change in social support from baseline to 6-months
  Family social support for healthy eating scale; 13 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from family - eating | Change in social support from baseline to 12-months
  Family social support for healthy eating scale; 13 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from family - eating | Change in social support from baseline to 24-months
  Family social support for healthy eating scale; 13 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from family - eating | Change in social support from baseline to 36-months
  Family social support for healthy eating scale; 13 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from friend - physical activity | Change in social support from baseline to 6-months
  Friend social support for physical activity scale; 9-items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from friend - physical activity | Change in social support from baseline to 12-months
  Friend social support for physical activity scale; 9-items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from friend - physical activity | Change in social support from baseline to 24-months
  Friend social support for physical activity scale; 9-items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from friend - physical activity | Change in social support from baseline to 36-months
  Friend social support for physical activity scale; 9-items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from family - physical activity | Change in social support from baseline to 6-months
  Family social support for physical activity scale; 15 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from family - physical activity | Change in social support from baseline to 12-months
  Family social support for physical activity scale; 15 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from family - physical activity | Change in social support from baseline to 24-months
  Family social support for physical activity scale; 15 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Social support from family - physical activity | Change in social support from baseline to 36-months
  Family social support for physical activity scale; 15 items using a 5-point Likert scale from None of the Time (1) to All of the Time (5) where a higher mean score indicated greater social support; Sallis et al., 1987
Outcome expectancies | Change in outcome expectancies from baseline to 6-months
  Outcome expectancies of behavior change; 25 items using 4-point Likert scale from Not True At All (1) to Exactly True (4); higher mean score indicating greater outcome expectancy; Huttunen-Lenz et al., 2018
Outcome expectancies | Change in outcome expectancies from baseline to 12-months
  Outcome expectancies of behavior change; 25 items using 4-point Likert scale from Not True At All (1) to Exactly True (4); higher mean score indicating greater outcome expectancy; Huttunen-Lenz et al., 2018
Outcome expectancies | Change in outcome expectancies from baseline to 24-months
  Outcome expectancies of behavior change; 25 items using 4-point Likert scale from Not True At All (1) to Exactly True (4); higher mean score indicating greater outcome expectancy; Huttunen-Lenz et al., 2018
Outcome expectancies | Change in outcome expectancies from baseline to 36-months
  Outcome expectancies of behavior change; 25 items using 4-point Likert scale from Not True At All (1) to Exactly True (4); higher mean score indicating greater outcome expectancy; Huttunen-Lenz et al., 2018
Coping self-efficacy | Change in coping self-efficacy from baseline to 6-months
  Coping self-efficacy scale; 14 items using a 4-point Likert scale from Not True At All (1) to Exactly True (4); higher mean score indicates greater self-efficacy for coping; Huttunen-Lenz et al., 2018
Coping self-efficacy | Change in coping self-efficacy from baseline to 12-months
  Coping self-efficacy scale; 14 items using a 4-point Likert scale from Not True At All (1) to Exactly True (4); higher mean score indicates greater self-efficacy for coping; Huttunen-Lenz et al., 2018
Coping self-efficacy | Change in coping self-efficacy from baseline to 24-months
  Coping self-efficacy scale; 14 items using a 4-point Likert scale from Not True At All (1) to Exactly True (4); higher mean score indicates greater self-efficacy for coping; Huttunen-Lenz et al., 2018
Coping self-efficacy | Change in coping self-efficacy from baseline to 36-months
  Coping self-efficacy scale; 14 items using a 4-point Likert scale from Not True At All (1) to Exactly True (4); higher mean score indicates greater self-efficacy for coping; Huttunen-Lenz et al., 2018

OTHER OUTCOMES:
Eligible DPP patients (reach) | Baseline to 3-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Eligible DPP patients (reach) | Baseline to 6-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Eligible DPP patients (reach) | Baseline to 9-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Eligible DPP patients (reach) | Baseline to 12-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Eligible DPP patients (reach) | Baseline to 15-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Eligible DPP patients (reach) | Baseline to 18-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Eligible DPP patients (reach) | Baseline to 21-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Eligible DPP patients (reach) | Baseline to 24-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Eligible DPP patients (reach) | Baseline to 27-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Eligible DPP patients (reach) | Baseline to 30-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Eligible DPP patients (reach) | Baseline to 33-months
  Proportion of patients eligible for DPP relative to total number of patients in ambulatory setting; electronic health record
Patients eligible for DPP (reach) | Baseline to 36-months
  Total number of patients in the ambulatory setting eligible for DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 3-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 6-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 9-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 12-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 15-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 18-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 21-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 24-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 27-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 30-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 33-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients referred to DPP (reach) | Baseline to 36-months
  Total number of patients in the ambulatory setting referred to DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 3-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 6-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 9-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 12-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 15-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 18-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 21-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 24-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 27-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 30-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 33-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Patients enrolled in DPP (reach) | Baseline to 36-months
  Total number of patients in the ambulatory setting enrolled in DPP; electronic health record
Referring clinical sites (adoption) | Baseline to 3-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 6-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 9-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 12-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 15-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 18-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 21-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 24-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 27-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 30-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 33-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring clinical sites (adoption) | Baseline to 36-months
  Total number of clinical sites referring patients to the DPP, electronic health record
Referring providers (adoption) | Baseline to 3-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 6-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 9-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 12-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 15-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 18-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 21-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 24-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 27-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 30-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 33-months
  Total number of providers referring patients to the DPP; electronic health record
Referring providers (adoption) | Baseline to 36-months
  Total number of providers referring patients to the DPP; electronic health record
Implementation | Continuous processual evaluation
  Qualitative assessment of implementation processes

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Gamble, PhD, MS, Principal Investigator — University of Mississippi Medical Center; Tamkeen Khan, PhD, Principal Investigator — American Medical Association
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gamble A, Khan T, Hughes A, Guo Y, Vasaitis S, Bidwell J, Christman B. Telehealth Diabetes Prevention Program for Adults With Prediabetes in an Academic Medical Center Setting: Protocol for a Hybrid Type III Trial. JMIR Res Protoc. 2023 Nov 13;12:e50183. doi: 10.2196/50183. PMID 37955955